CLINICAL TRIAL: NCT02074917
Title: Comparison of Dynamic Knee Stability and Functional Outcomes in Anatomical Single-bundle ACL at Anteromedial or Central Tunnel Position - Prospective, Randomized and Double-blind Clinical Trial in Athletes
Brief Title: Comparison of Dynamic Knee Stability and Functional Outcomes in Anatomical ACL Reconstruction at AM or Central Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Arnaldo José Hernandez, Associate Professor, PhD, MSc, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCFMUSP972
Record Dates: First submitted 2013-10-24; First posted 2014-02-28 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Rupture of Anterior Cruciate Ligament; Complete Tear, Knee, Anterior Cruciate Ligament
Keywords: anterior cruciate ligament; ACL; anterior cruciate ligament reconstruction; outcome assessment; outcome assessment, patient; treatment outcome; exercise test; anatomic; anatomical; single-bundle; force platform; postural balance; biomechanics; CT scan; X-ray computed tomography; tomography; diagnostic imaging; knee; knee injuries; joint instability; reconstructive surgical procedures; knee surgery; arthroscopy; athletes; sports medicine; humans; prospective studies; Randomized Controlled Trial
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries; Joint Instability | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AM anatomical ACL reconstruction (Experimental): Femoral and tibial tunnels performed in anteromedial footprint of ACL reconstruction
  Interventions: Procedure: Anatomical ACL reconstruction
- CENTRAL anatomical ACL reconstruction (Experimental): Femoral and tibial tunnels performed in the center of ACL footprint
  Interventions: Procedure: Anatomical ACL reconstruction

INTERVENTIONS:
Procedure: Anatomical ACL reconstruction — Anatomical anterior cruciate ligament reconstruction in the anteromedial or central tunnels positions.
  Other Names: anatomic ACL reconstruction; anatomic anterior cruciate ligament reconstruction; anatomical anterior cruciate ligament reconstruction; anterior cruciate ligament reconstruction; anterior cruciate ligament; ACL

SUMMARY:
This is a prospective, randomized and double-blind clinical trial about anatomical single-bundle anterior cruciate ligament (ACL) reconstruction.

One of the most common causes of ACL reconstruction failure is poor graft positioning. There is evidence that graft placement aligned with native insertion sites results in superior clinical outcomes. Current anatomic ACL reconstruction concepts highlight the importance of the native anatomy to restore physiological knee kinematics more accurately.

This study aims to investigate clinical outcomes and dynamic knee stability with force platform and other functional tests after ACL reconstruction in two different groups of tunnel position: anteromedial ACL footprint (AM) or central ACL footprint.

It was hypothesized that there would be clinical or dynamic stability differences between AM or Central tunnel groups in ACL reconstruction.

DETAILED DESCRIPTION:
Tunnel position will be recorded and confirmed with postoperative computer tomography.

ELIGIBILITY:
Inclusion Criteria:

* Physical activity classified by Tegner scale ≥ 5
* Absence of other associated ligament injuries in the operated knee
* No ACL rerupture or previous ACL reconstruction in the same or other knee
* Absence of untreated lesions of the opposite knee
* No obvious change in the alignment of the mechanical axis that required surgical correction
* Athletes of both gender with a minimum age of 18 years and maximum of 45 years
* Signature of the consent term (IRB)
* Not be pregnant.

Exclusion Criteria:

* Request to stop the study by patient at any time
* Fracture not associated with the surgical procedure
* Do not carry out the rehabilitation protocol as oriented by the Sports Medicine group.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Dynamic Stability with force platform | 12 months
  Evaluation of dynamic stability in stand position and leg movements with force platform

SECONDARY OUTCOMES:
Change from baseline and between groups in Lysholm knee scoring scale | 6, 12, 24 months
  This is a validated scoring scale to evaluate outcomes of knee ligament surgery, particularly symptoms of instability. The total score is the sum of each response to the 8 items, of a possible score of 100.
Change from baseline and between groups in Tegner activity score | 6, 12, 24 months
  This is a validated score for level of activity related to knee stability. It provides a standardized method of grading work and sporting activities from 0 to 10.
Single leg hop test for distance - side to side difference | 6, 12 months
  This test includes a single leg hop for distance comparison between involved leg vs. contra-lateral normal leg. Results are expressed as a percentage of the non-involved leg.
Isokinetic knee strength test - side to side difference | 6, 12 months
  Quadriceps and hamstring isokinetic strength are assessed at velocities of 60 and 240 degrees per second and values are compared between involved operated leg and non-involved leg and between groups. Peak torque and flexion/extension rate are analyzed.
Change from baseline and between groups in Dynamic Stability with force platform | 6 months
  Evaluation of dynamic stability in stand position and leg movements with force platform. Antero-posterior and latero-medial movements are measured in metric scale. Area and velocity of movement are also calculated.
Change from baseline and between groups in International Knee Documentation Committee form (IKDC) | 6, 12 e 24 months
  The form is used to detect improvement or deterioration in symptoms, function, and sports activities due to knee impairment. It is a validated 18-item patient measurement tool. that can be used for post-operatory ACL reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Arnaldo J Hernandez, PhD, MSc, MD, Principal Investigator — University of Sao Paulo; Danilo RO Oliveira, MD, Study Director — University of Sao Paulo; Tiago L Fernandes, MSc, MD, Study Director — University of Sao Paulo; Ellen CR Felix, Study Director — University of Sao Paulo
Locations (1):
- Instituto de Ortopedia e Traumatologia do HCFMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Zantop T, Wellmann M, Fu FH, Petersen W. Tunnel positioning of anteromedial and posterolateral bundles in anatomic anterior cruciate ligament reconstruction: anatomic and radiographic findings. Am J Sports Med. 2008 Jan;36(1):65-72. doi: 10.1177/0363546507308361. Epub 2007 Oct 11. PMID 17932407
- [Background] Misonoo G, Kanamori A, Ida H, Miyakawa S, Ochiai N. Evaluation of tibial rotational stability of single-bundle vs. anatomical double-bundle anterior cruciate ligament reconstruction during a high-demand activity - a quasi-randomized trial. Knee. 2012 Mar;19(2):87-93. doi: 10.1016/j.knee.2011.01.003. Epub 2011 Feb 12. PMID 21316972
- [Background] Forsythe B, Kopf S, Wong AK, Martins CA, Anderst W, Tashman S, Fu FH. The location of femoral and tibial tunnels in anatomic double-bundle anterior cruciate ligament reconstruction analyzed by three-dimensional computed tomography models. J Bone Joint Surg Am. 2010 Jun;92(6):1418-26. doi: 10.2106/JBJS.I.00654. PMID 20516317
- [Background] Musahl V, Plakseychuk A, VanScyoc A, Sasaki T, Debski RE, McMahon PJ, Fu FH. Varying femoral tunnels between the anatomical footprint and isometric positions: effect on kinematics of the anterior cruciate ligament-reconstructed knee. Am J Sports Med. 2005 May;33(5):712-8. doi: 10.1177/0363546504271747. Epub 2005 Feb 16. PMID 15722268
- [Background] Mohammadi F, Salavati M, Akhbari B, Mazaheri M, Khorrami M, Negahban H. Static and dynamic postural control in competitive athletes after anterior cruciate ligament reconstruction and controls. Knee Surg Sports Traumatol Arthrosc. 2012 Aug;20(8):1603-10. doi: 10.1007/s00167-011-1806-4. Epub 2011 Nov 29. PMID 22124847